CLINICAL TRIAL: NCT02512484
Title: Improving the Detection of Active Tuberculosis in Accident and Emergency (A&E) Departments
Brief Title: Improving the Detection of Active Tuberculosis in Accident and Emergency Departments
Acronym: ACE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Public Health England (Other Government)
Responsible Party: Principal Investigator, Jo Southern, Clinical Research Lead, Public Health England
Other Study IDs: TB A&E study
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Latent Tuberculosis; Active Tuberculosis
Keywords: tuberculosis; accident and emergency
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis; Emergencies | interventions — Blood Specimen Collection; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retention of residual blood samples after inital testing, with appropriate consent to do so from individuals and ethics committee.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- high risk TB individuals attending A&E Departments: Assessment against inclusion/exclusion criteria in terms of risk of TB. If eligible, assessment and testing as appropriate for active or latent TB
  Interventions: Procedure: venepuncture, sputum collection, xray

INTERVENTIONS:
Procedure: venepuncture, sputum collection, xray — venepuncture, sputum collection, xray

SUMMARY:
Tuberculosis (TB) control remains a public health challenge. Many people in the UK do not have a general practitioner (GP) registration and their only interaction with the NHS is via Accident and Emergency (A&E) Departments of hospitals. This is often the case for those in hard to reach groups, who are also those often at highest risk of TB. This study seeks to assess whether A&E Departments are effective sites for the identification and onward management of TB, both in its latent and active forms.

DETAILED DESCRIPTION:
This proposal is focused upon early diagnosis, referral and treatment of active tuberculosis, which has two key components: 1) ensuring optimal outcome for individuals; 2) contributing to disease control in public health terms by preventing further spread.

A&E Departments are an important point of testing and referral for the client group that constitute those at greatest risk, as for many this will be their only interaction with the health service. Currently, A&E Departments contribute about 20% of those diagnosed with TB. The majority of these individuals are most likely to have presented with symptoms indicative of disease, compared to those attending for other reasons who would have been unlikely to have been tested or referred.

This study will seek to evaluate specific measures currently being undertaken by Public Health England and the NHS to control TB as well as investigate whether case finding for active TB in A&E departments would improve TB control. The economic impact of these interventions will be evaluated, providing a measure of its value for money.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 16 years or older, who are new entrants from high incidence countries who have arrived in the UK within the past 2 years or those born in high incidence countries who entered the UK more than five years ago, but have spent more than one year (cumulative) in the past five years in a high incidence country.
2. Those with social risk factors who have signs and/or symptoms of TB.

Exclusion Criteria:

1. Individuals who are under 16 years
2. Individuals who were born in the UK or a low incidence countries and do not have risk factors

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals at high risk of TB
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
xray diagnosis of active TB | 1 year
  clinical signs and symptoms on xray

SECONDARY OUTCOMES:
diagnosis of latent TB | 1 year
  positive blood test result by interferon gamma release assay (IGRA) in line with the manufacturer instructons for the test

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Barts NHS Trust, London, London
  - Ealing Hospital, London, London
  - West Middlesex Hospital NHS Trust, London, London

REFERENCES:
- [Derived] Gupta RK, Lule SA, Krutikov M, Gosce L, Green N, Southern J, Imran A, Aldridge RW, Kunst H, Lipman M, Lynn W, Burgess H, Rahman A, Menezes D, Rahman A, Tiberi S, White PJ, Abubakar I. Screening for tuberculosis among high-risk groups attending London emergency departments: a prospective observational study. Eur Respir J. 2021 Jun 24;57(6):2003831. doi: 10.1183/13993003.03831-2020. Print 2021 Jun. PMID 33737408